CLINICAL TRIAL: NCT00605774
Title: Hypoglycemia Associated Autonomic Failure in Type 1 DM, Question 5
Brief Title: Hypoglycemia Associated Autonomic Failure in Type 1 DM, Q5
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Steve Davis, Chairman of Medicine, University of Maryland, Baltimore, Vanderbilt University
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: IRB #040911- HAAF in T1DM, Q5; R01DK069803-03 (NIH)
Record Dates: First submitted 2008-01-18; First posted 2008-01-31 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Type 1 Diabetes
Keywords: catecholamines; diabetes; exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Motor Activity | interventions — Epinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Hyperinsulinemic euglycemic glucose clamps x 2 on Day 1 Hyperinsulinemic euglycemic glucose clamp with epinephrine infusion on Day 2
  Interventions: Drug: epinephrine
- 2 (Experimental): Day 1 euglycemic exercise period x 2 Day 2 hyperinsulinemic euglycemic glucose clamp with epinephrine infusion
  Interventions: Drug: epinephrine

INTERVENTIONS:
Drug: epinephrine — Epinephrine 0.06 µg/kg/min infused over two hours during experimental period on Day 2
  Arms: 1
Drug: epinephrine — Epinephrine 0.06 µg/kg/min infusion during hyperinsulinemic euglycemic clamp on day 2
  Arms: 2

SUMMARY:
When a patient with Type 1 diabetes exercises, he or she is more prone to low blood sugar, or hypoglycemia. It is known that antecedent exercise can blunt defense responses, called counterregulatory responses to subsequent hypoglycemia in Type 1 DM, causing him or her to be vulnerable to another bout of hypoglycemia. Epinephrine is one of the important hormones in the defense of blood glucose during both exercise and hypoglycemia. We will test the hypothesis that antecedent exercise will blunt the metabolic, neuroendocrine and cardiovascular effects of subsequent epinephrine infusion in Type 1 DM.

DETAILED DESCRIPTION:
We have recently performed studies to determine whether the critical metabolic actions of epinephrine are blunted in Type 1 DM. These studies have obvious clinical relevance because strategies aimed at increasing circulating levels of epinephrine will not be effective if the metabolic counterregulatory mechanisms (increased endogenous glucose production (EGP), increased lipolysis and reduced glucose uptake) of the hormone are also blunted. Epinephrine was infused to reach circulating levels of ~ 1000 pg/ml (This level of epinephrine is equivalent to values of the hormone observed during hypoglycemia of 50 mg/dl in healthy males and T1DM men with average glucose control) in groups of either intensively treated (HBA1C < 7.0%), conventionally treated (HBA1C > 9.0%) type 1 DM and age, weight matched healthy controls. In the intensively treated DM group, epinephrine's actions to increase EGP, lipolysis and to restrain glucose uptake were significantly reduced (<60%). The mechanism for our finding needs to be determined. Our hypothesis is that antecedent exercise can cause repetitive activations of Autonomic-adrenomedullary responses that lead to downregulation of β-adrenoreceptor mechanisms. Therefore, the combination of blunted epinephrine effects, increased insulin action and reduced levels of the catecholamine might fully explain the vexing clinical question of post exercise hypoglycemia in Type 1 DM. In this application, we will test the hypothesis that antecedent exercise will blunt the metabolic, neuroendocrine and cardiovascular effects of subsequent epinephrine infusion in Type 1 DM.

ELIGIBILITY:
Inclusion Criteria:

* 28 (14 males, 14 females) conventionally treated Type 1 diabetic patients with HA1C > 8.5%
* 28 (14 males, 14 females) intensively treated Type 1 diabetic patients with HA1C < 7%
* 28 (14 males, 14 females) non-diabetic controls
* Age 18-45 yr.
* Had diabetes for 2-15 years if diabetic subject
* No clinical evidence of diabetic tissue complications, no cardiovascular disease
* Body mass index 21-27kg · m-2
* Normal bedside autonomic function
* Normal results of routine blood test to screen for hepatic, renal, and hematological abnormalities
* Female volunteers of childbearing potential: negative HCG pregnancy test

Exclusion Criteria:

* Prior history of poor health: any current or prior disease condition that alters carbohydrate metabolism and prior cardiac events and/or evidence for cardiac disease
* Hemoglobin of less than 12 g/dl
* Abnormal results following screening tests
* Pregnancy
* Subjects unable to give voluntary informed consent
* Subjects with a recent medical illness
* Subjects with known liver or kidney disease
* Subjects taking steroids
* Subjects taking beta blockers
* Subjects on anticoagulant drugs, anemic, or with known bleeding diseases

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
catecholamine levels | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Stephen N. Davis, MD, Principal Investigator — Vanderbilt University